CLINICAL TRIAL: NCT02212028
Title: Pharmacodynamic and Pharmacokinetic Profiles of Prasugrel in Patients With ST Elevation Myocardial Infarction: A Randomized Comparison of Standard Versus Crushed Formulation
Brief Title: Pharmacological Effects of Crushing Prasugrel in STEMI Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prasugrel-CRUSH
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Results first posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2015-08

CONDITIONS: Coronary Artery Disease
Keywords: ST-elevation myocardial infarction; prasugrel; pharmacodynamic; pharmacokinetic
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction | interventions — Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prasugrel crush (Experimental): Prasugrel 60mg loading dose as crushed tablets
  Interventions: Drug: prasugrel
- Prasugrel tablets (Active Comparator): Prasugrel 60 mg loading dose as whole tablets
  Interventions: Drug: prasugrel

INTERVENTIONS:
Drug: prasugrel — the effects of whole tablets versus crushed tablets will be compared
  Other Names: Effient

SUMMARY:
Prasugrel has shown to be superior to clopidogrel, in adjunct to aspirin, in preventing recurrent ischemic events. Prasugrel is approved in patients with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) at a dosage of 60 mg loading dose (LD) followed by 10 mg/day. However, a delay in the onset of its antiplatelet effects in this particular setting has been consistently shown. administration of clopidogrel and ticagrelor crushed tablets has been tested and a faster and greater bioavailability compared to the whole tablets has been observed. However, if the administration of a crushed prasugrel LD may overcome the above limitation is still unknown and represents the aim of our study. The proposed investigation will have a prospective, randomized, design in which STEMI patients undergoing primary PCI will be randomized to receive two different formulation of prasugrel LD (60 mg whole tablets and 60 mg crushed tablets). Pharmacodynamic testing will be performed at several time points to test our study hypothesis that crushed LD regiment will achieve more prompt and enhanced platelet inhibitory effects.

DETAILED DESCRIPTION:
Dual antiplatelet therapy consisting of aspirin and a P2Y12 receptor antagonist is the cornerstone of treatment for prevention of thrombotic events in patients with acute coronary syndromes (ACS). Prasugrel, a third generation thienopyridine, is an orally administered prodrug that needs single-step hepatic biotransformation into its active metabolite to irreversibly block the P2Y12 receptor. Prasugrel has shown to be superior to clopidogrel, in adjunct to aspirin, in preventing recurrent ischemic events. Prasugrel is approved in patients with ST-elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI) at a dosage of 60 mg loading dose (LD) followed by 10 mg/day. However, a delay in the onset of its antiplatelet effects in this particular setting has been consistently shown. The STEMI setting is characterized by conditions, such as impaired absorption and hepatic metabolism, patients either intubated, in shock or unable to swallow, which may affect the pharmacoki¬netic and pharmacodynamic effects of orally administered antiplatelet drugs. The administration of clopidogrel and ticagrelor crushed tablets has been tested and a faster and greater bioavailability compared to the whole tablets has been observed. However, if the administration of a crushed prasugrel LD may overcome the above limitation is still unknown and represents the aim of our study. The proposed investigation will have a prospective, randomized, design in which STEMI patients undergoing primary PCI will be randomized to receive two different formulation of prasugrel LD (60 mg whole tablets and 60 mg crushed tablets). Pharmacodynamic testing will be performed at several time points to test our study hypothesis that crushed LD regiment will achieve more prompt and enhanced platelet inhibitory effects. This study will provide insights on the pharmacodynamic effects of crushed prasugrel LD and will help clinicians choose the most appropriate treatment to avoid complications related to inadequate platelet inhibition in the early phase of patients with STEMI undergoing primary PCI.

ELIGIBILITY:
Inclusion criteria:

* Patients with ST-elevation myocardial infarction undergoing primary PCI
* Age between 18 and 75 years old

Exclusion criteria:

* Age >75 years
* Weight <60 Kg
* On treatment with a P2Y12 receptor antagonist (ticlopidine, clopidogrel, prasugrel, ticagrelor) in past 7 days
* Known allergies to aspirin or prasugrel
* Considered at high risk for bleeding
* History of ischemic or hemorrhagic stroke or transient ischemic attack
* On treatment with oral anticoagulant (Vitamin K antagonists, dabigatran, rivaroxaban, apixaban)
* Treatment with IIb/IIIa glycoprotein inhibitors
* Fibrinolytics within 24 hours
* Known blood dyscrasia or bleeding diathesis
* Known platelet count <80x106/mL
* Known hemoglobin <10 g/dL
* Active bleeding
* Hemodynamic instability
* Known creatinine clearance <30 mL/minute
* Known severe hepatic dysfunction
* Pregnant females*

  * Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick Angiolillo, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rollini F, Franchi F, Hu J, Kureti M, Aggarwal N, Durairaj A, Park Y, Seawell M, Cox-Alomar P, Zenni MM, Guzman LA, Suryadevara S, Antoun P, Bass TA, Angiolillo DJ. Crushed Prasugrel Tablets in Patients With STEMI Undergoing Primary Percutaneous Coronary Intervention: The CRUSH Study. J Am Coll Cardiol. 2016 May 3;67(17):1994-2004. doi: 10.1016/j.jacc.2016.02.045. Epub 2016 Mar 21. PMID 27012781

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between October 15, 2014, and August 12, 2015, there were a total of 123 patients presenting with a STEMI at the University of Florida Health-Jacksonville, that were screened.
Pre-assignment Details: 45 patients did not meet study entry criteria, while 78 provided their written informed consent to participate in the study and, of these, 52 were randomized. the remaining subjects were not randomized because of exclusion criteria emerged after consenting.
Groups:
- Prasugrel Tablets: Prasugrel 60 mg loading dose whole tablets
Period: Overall Study
Arm/Group | Prasugrel Crush | Prasugrel Tablets
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Two patients in the whole tablets arm were excluded from the analysis because of missing data for the primary end point.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel Crush | Prasugrel Tablets | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9) | 58 (10) | 58 (10)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 19 | 18 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units (PRU)
Description: The primary end-point of the study is the comparison in platelet reactivity expressed as PRU determined by VerifyNow P2Y12 between prasugrel 60 mg and crushed prasugrel 60 mg at 2 hours after LD administration
Time Frame: 2 hrs
Population: The primary population was defined as patients who received the randomized treatment and had a valid primary end point value (PRU at 2 hours) and was considered for analysis of all endpoints.
Measure: Least Squares Mean (95% Confidence Interval); unit: PRU
Arm/Group | Prasugrel Crush | Prasugrel Tablets
Number analyzed (Participants) | 26 | 24
PRU | 95 [55 to 135] | 164 [122 to 206]
Statistical Analysis 1: Comparison: Prasugrel Crush; Test type: Superiority or Other; p = 0.022, ANOVA; Mean Difference (Final Values) = 68, 95% CI 2-sided [10 to 126]

2. Secondary Outcome: Platelet Reactivity Index (PRI)
Description: The secondary end-point of the study is the comparison in platelet reactivity expressed as PRI determined by whole blood vasodilator-stimulated phosphoprotein (VASP) between prasugrel 60 mg and crushed prasugrel 60 mg at 2 hours after LD administration
Time Frame: 2 hrs
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: PRI
Arm/Group | Prasugrel Crush | Prasugrel Tablets
Number analyzed (Participants) | 26 | 24
PRI | 33 [20 to 46] | 61 [47 to 75]
Statistical Analysis 1: Comparison: Prasugrel Crush vs Prasugrel Tablets; Test type: Superiority or Other; p = 0.005, ANOVA

ADVERSE EVENTS:
Time Frame: 3 days
Description: In-hospital adverse events, including ischemic and bleeding complications were recorded.
Arm/Group | Prasugrel Crush | Prasugrel Tablets
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 1/26 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Crush (N=26) | Prasugrel Tablets (N=26)
Minor bleeding (Renal and urinary disorders) | 1 (1) | 0 (0) — There was only 1 minor bleeding event (hematuria) in the crushed prasugrel arm, which did not required drug discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes